CLINICAL TRIAL: NCT00116441
Title: Vaccination in the Peripheral Stem Cell Transplant Setting for Multiple Myeloma: The Use of Autologous Tumor Cells With an Allogeneic GM-CSF Producing Cell Line
Brief Title: Vaccination in the Peripheral Stem Cell Transplant Setting for Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-0007; K-0007
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; PSCT; Peripheral Stem Cell Transplant; Chemotherapy; GVAX
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

INTERVENTIONS:
Biological: Therapeutic Cellular Vaccine, GM-CSF Producing

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of vaccination with autologous myeloma cells and an allogeneic granulocyte-macrophage colony stimulating factor (GM-CSF) producing cell line.

ELIGIBILITY:
Inclusion Criteria:

* De novo multiple myeloma
* ECOG 0-2
* No serious co-morbid illnesses and adequate organ function
* > 4 weeks from systemic steroids

Exclusion Criteria:

* No existing secondary malignancies and no history of secondary malignancies in the past 5 years
* No active autoimmune disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2000-10; Study Completion 2004-10

PRIMARY OUTCOMES:
Multiple myeloma

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States